CLINICAL TRIAL: NCT03106376
Title: Magnetic Resonance Spectroscopy Studies of Acute Hypoxic and Hyperoxic Breathing in Healthy Volunteers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study team has decided to focus on other projects
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Dost Ongur, Professor of Psychiatry, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017P000328
Record Dates: First submitted 2017-03-29; First posted 2017-04-10 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Experimental): 16% O2 gas in breathed air for 30 minutes 26% O2 gas in breathed air for 30 minutes
  Interventions: Other: 16% O2 gas in breathed air; Other: 26% O2 gas in breathed air

INTERVENTIONS:
Other: 16% O2 gas in breathed air — Inspiratory gas mixtures: Hypoxic inspiratory gas will be obtained by adding nitrogen (N2) to normobaric, normoxic air with medical N2 tanks.
  Delivery of gas mixture: The gas mixture will be delivered by standard tight facemask.
Other: 26% O2 gas in breathed air — Inspiratory gas mixtures: Hyperoxic inspiratory gas will be obtained by adding oxygen (O2) to normobaric, normoxic air with medical O2 tanks.
  Delivery of gas mixture: The gas mixture will be delivered by standard tight facemask.

SUMMARY:
This study evaluates the impact of hypoxic and hyperoxic breathing on measures of brain redox balance and metabolism in healthy individuals. All participants will undergo an MRI scan during administration of air mixtures with different oxygen concentrations to collect the brain measures.

DETAILED DESCRIPTION:
Molecular oxygen (O2) constitutes 21% of the air people breathe at sea level. But humans can safely be exposed to somewhat lower and higher concentrations of oxygen. The varying amounts of oxygen entering the body modulate the oxygen available in tissue, ultimately leading to change in redox balance and metabolism. The investigators recently developed non-invasive MRI-based techniques to quantify redox balance and ATP generation in the brain. These processes are thought to be abnormal in people with psychiatric disorders.

In this study, the investigators aim to manipulate the concentration of oxygen in the breathed air in 2 separate MRI scans on consecutive days (16% and 26%). The investigators anticipate that healthy individuals will demonstrate changes in brain redox balance and metabolism in response to these modulations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals age between 18 and 40 years old
* BMI between 19 and 29 kg/m2
* Having capacity to consent to the study

Exclusion Criteria:

* Under 18 or over 40 Family history of psychiatric illness among first degree relatives (parents, siblings, or children)
* Delirium secondary to medical illness
* Any contraindication to MR scan, including claustrophobia, pregnancy, etc.
* Medical condition that might endanger the subject during or after a blood draw (e.g. hemophilia)
* Significant medical or neurological illness
* Prior high altitude pulmonary edema (HAPE) or high-altitude cerebral edema (HACE) diagnosis Born at altitudes greater than 2,100 m (~7,000 ft) Systemic disease with or without any functional limitation; including controlled hypertension controlled diabetes without systemic effects any cardiac conditions with or without functional limitation, such as, coronary artery disease or valve disease Pregnancy determined by urine pregnancy test, detecting presence of human chorionic gonadotropin (hCG), less than six weeks postpartum, or planning to conceive during the study period.

Women who are not willing to receive serum pregnancy tests Active smoking and tobacco chewers. Volunteers may be enrolled if they quit smoking for more than 1 year.

Excess alcohol use: more than ½ L/day of wine consumption or equivalent Any current medication use except oral contraceptives. Living in areas that are more than 1,200 m (~4,000 feet), or have traveled to areas that are more than 1,200 m for more than four days within the last 2 months Anemia, as defined by hemoglobin < 10g/dL Abnormal hemoglobin (e.g. presence of hemoglobin S) Evidence of apnea or other sleeping disorders Evidence of asthma Lower respiratory infection within the last 30 days Not willing to have blood drawn from an arm vein each test day of the study Claustrophobia (inability to tolerate MRI scan or wear a facemask) Currently enrolled in another research study Facial abnormalities that would preclude proper use of a face mask Hb<12

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-29 (Estimated); Primary Completion 2023-08-29 (Estimated); Study Completion 2023-08-29 (Estimated)

PRIMARY OUTCOMES:
NAD+/NADH ratio | During 30 minute hypoxic/hyperoxic exposure portion of the MRS scan
  NAD+ and NADH concentrations are measured using 31P MRS scanning

SECONDARY OUTCOMES:
CK Kf | During 30 minute hypoxic/hyperoxic exposure portion of the MRS scan
  Reaction rate of the creatine kinase enzyme measured using 31P MRS scanning
PCr | During 30 minute hypoxic/hyperoxic exposure portion of the MRS scan
  Phosphocreatine concentration measured using 31P MRS scanning
Pi | During 30 minute hypoxic/hyperoxic exposure portion of the MRS scan
  Inorganic phosphate concentration measured using 31P MRS scanning
ATP | During 30 minute hypoxic/hyperoxic exposure portion of theMRS scan
  ATP concentration measured using 31P MRS scanning

CONTACTS AND LOCATIONS:
Overall Officials: Dost Ongur, MD PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No